CLINICAL TRIAL: NCT04800302
Title: Ultrasound-guided Continuous Quadratus Lumborum Block III for Postoperative Analgesia in Percutaneous Nephrolithotomy
Brief Title: U/S-guided Continuous Quadratus Lumborum Block III in Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: USGCQLBIIIPCNL
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Analgesia; Surgery; Renal Stone
Keywords: Quadratus Lumborum Block III; Ultrasound-guided; Percutaneous nephrolithotomy; Analgesia
MeSH Terms: conditions — Agnosia; Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous QLB group (Experimental): U/S-guided continous QLB III
  Interventions: Procedure: Continous Quadratum Lumborum Block III; Procedure: Single dose Quadratum Lumborum Block III; Procedure: Intra-venous Morphine
- Single dose QLB group (Active Comparator): U/S-guided single dose QLB III
  Interventions: Procedure: Single dose Quadratum Lumborum Block III; Procedure: Intra-venous Morphine
- Morphine group (Active Comparator): IV Morphine
  Interventions: Procedure: Intra-venous Morphine

INTERVENTIONS:
Procedure: Continous Quadratum Lumborum Block III — Continuous infusion of Bupivacaine 0.125 % at a rate of 0.1 ml/kg/hr (not exceeding 12 ml/hour), infused through a catheter inserted in the plane between quadratus lumborum & psoas major muscles with ultrasound guidance.
  Arms: Continuous QLB group
Procedure: Single dose Quadratum Lumborum Block III — Single injection of a mixture solution of 20 ml Bupivacaine 0.5% + 10 ml Lidocaine 2%, injected through a needle inserted at the posterior aspect of the quadratus lumborum muscle between it and erector spinae muscle with ultrasound guidance.
  Arms: Continuous QLB group; Single dose QLB group
Procedure: Intra-venous Morphine — Intra-venous Morphine [0.1 mg/kg] as rescue analgesic shots when the Visual Analogue Score (VAS) for pain exceeds 4.

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is considered to be the first choice and a more conservative procedure than open stone surgery. Not only postoperative pain related to dilatation of the renal capsule and parenchymal tract, but also patient's discomfort & nephrostomy tube-related stress are reported to delay recovery time and increase the complication rates. This study is designed to provide postoperative analgesia by using ultrasound-guided continuous Quadratus Lumborum Block (QLB) III in patients undergoing PCNL and to assess pain scores & side effects with less opioids consumption.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II.
* Scheduled for percutaneous nephrolithotomy (PCNL).

Exclusion Criteria:

* Patient refusal.
* Coagulation disorders.
* Skin lesions or infection at site of needle insertion.
* Known allergy to local anesthetics or opioids.
* Patients suffering from neurological or mental disease.
* Procedure turned into open stone surgery.
* Failure of identification by U/S.
* Urinary tract malignancies.
* Opioid consumption 48 hours before the operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Morphine consumption. | 24 hours
  Total dose of Morphine (measured in mg) given intra-venously to the patient post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif A Embaby, MSc, Principal Investigator — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided